CLINICAL TRIAL: NCT06995404
Title: Transversus Abdominis Plane Block (TAP) Versus Thoracoabdominal Nerve Block Through Perichondrial Approach (M-TAPA) in Laparoscopic Gynecologic Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ela Erdem Hıdiroglu, MD, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AESH-EK-2025-028
Record Dates: First submitted 2025-04-28; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Gynecologic Laparoscopic Surgery; Regional Anesthesia Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (No Intervention)
- group TAP (Active Comparator)
  Interventions: Procedure: TAP Block Group
- group M-TAPA (Active Comparator)
  Interventions: Procedure: M-TAPA Block group

INTERVENTIONS:
Procedure: TAP Block Group — Patients in the TAP group will receive a bilateral Transversus Abdominis Plane (TAP) block under ultrasound guidance prior to surgery after general anaesthesia, with the local anesthetic administered between the internal oblique and transversus abdominis muscles. A total of 40 mL of 0.25% bupivacaine will be used for the procedure.
  Arms: group TAP
Procedure: M-TAPA Block group — Patients in the M-TAPA group will receive a bilateral Thoracoabdominal Nerve Block through Perichondrial Approach (M-TAPA) under ultrasound guidance prior to surgery after general anaesthesia. A total of 40 mL of 0.25% bupivacaine will be used for the procedure.
  Arms: group M-TAPA

SUMMARY:
Although laparoscopic techniques are considered minimally invasive surgical procedures with lower perioperative pain scores compared to open surgeries, they are still associated with significant levels of pain. This study aims to investigate the analgesic effectiveness of two routinely performed regional analgesic techniques in our clinic-ultrasound-guided classic bilateral TAP block and ultrasound-guided bilateral M-TAPA block-in patients undergoing laparoscopic gyneco-oncologic surgery (LGOS), as well as their effects on intraoperative opioid consumption.

ELIGIBILITY:
Inclusion Criteria:Female patients aged between 18 and 80 years, classified as ASA physical status I to III, undergoing laparoscopic gynecologic surgery under general anesthesia -

Exclusion Criteria:Coagulopathy

Neuropathy

Chronic analgesic therapy

Severe cardiopulmonary disease

Uncontrolled diabetes mellitus (HbA1c > 8%)

Severe renal or hepatic failure

Pregnancy or lactation

Body mass index (BMI) greater than 35 kg/m²

Local infection at the injection site

Inability to comprehend pain scores or cooperate (e.g., Alzheimer's disease, mental retardation)

Allergy to local anesthetic agents

Refusal to participate in the study

-

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 90 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of intraoperative opioid consumption | during surgery

SECONDARY OUTCOMES:
Comparison of postoperative Visual Analog Scale (VAS) pain scores | postoperative first day
  VAS is an eleven-scale pain score scored from 0 to 10, with vas 0 being no pain and vas 10 being maximum pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No